CLINICAL TRIAL: NCT02383589
Title: A Randomized, Double-Blind, Double-Dummy, Active-Comparator, Multicenter Study to Evaluate the Efficacy and Safety of Rituximab Versus MMF in Patients With Pemphigus Vulgaris
Brief Title: A Study to Evaluate the Efficacy and Safety of Rituximab Versus Mycophenolate Mofetil (MMF) in Participants With Pemphigus Vulgaris (PV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA29330; 2014-000382-41 (EudraCT Number)
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus | interventions — Mycophenolic Acid; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Mycophenolate Mofetil (MMF) (Active Comparator): Participants will receive MMF orally twice daily (every 12 hours, Q12H) from Day 1 to Week 52. Participants will also receive rituximab matching placebo by intravenous (IV) infusion on Days 1 and 15 with repeat administration on Days 168 and 182 provided specific safety criteria have been met.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Rituximab Placebo
- Rituximab (RTX) (Experimental): Participants will receive rituximab by IV infusion on Days 1 and 15 with repeat administration on Days 168 and 182 provided specific safety criteria have been met. Participants will also receive MMF matching placebo orally twice daily Q12H from Day 1 to Week 52.
  Interventions: Drug: Mycophenolate Mofetil Placebo; Drug: Rituximab

INTERVENTIONS:
Drug: Mycophenolate Mofetil Placebo — MMF matching placebo will be administered orally Q12H.
  Arms: Rituximab (RTX)
Drug: Mycophenolate Mofetil — MMF will be administered at a starting dose of 500 milligrams (mg) Q12H and the dose will be titrated to achieve a goal of 1 gram (gm) Q12H.
  Other Names: MMF, CellCept
  Arms: Mycophenolate Mofetil (MMF)
Drug: Rituximab — Rituximab will be administered at a dose of 1000 mg via IV infusion.
  Other Names: MabThera/Rituxan
  Arms: Rituximab (RTX)
Drug: Rituximab Placebo — Rituximab matching placebo will be administered via IV infusion.
  Other Names: MabThera/Rituxan
  Arms: Mycophenolate Mofetil (MMF)

SUMMARY:
This is a Phase III, randomized, double-blind, double-dummy, active-comparator, parallel-arm, multicenter study to evaluate the efficacy and safety of rituximab compared with MMF in participants with moderate-to-severely active PV requiring 60-120 milligrams per day (mg/day) oral prednisone or equivalent. Participants must have a confirmed diagnosis of PV within the previous 24 months (by skin or mucosal biopsy and immunohistochemistry) and evidence of active disease at screening.

Approximately 135 participants will be enrolled at up to 60 centers worldwide. Participants will be randomized in a 1:1 ratio to receive either rituximab plus MMF placebo or rituximab placebo plus MMF. Randomization will be stratified by duration of illness.

The study will consist of three periods: a screening period of up to 28 days, a 52-week double-blind treatment period, and a 48-week safety follow up period that begins at the time of study treatment completion or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PV within the previous 24 months, based on the presence of histological features of acantholysis via skin or mucosal biopsy and one of the following: tissue bound immunoglobulin G (IgG) antibodies by direct immunofluorescence on the surface of affected epithelium or serological detection of serum desmoglein-3 (DSg3) autoantibodies against epithelial cell surface either by indirect immunofluorescence microscopy or by enzyme-linked immunosorbent assay
* Presence of moderate-to-severely active disease, defined as overall PDAI activity score of greater than or equal to (>/=)15
* Receiving standard-of-care corticosteroids consisting of 60-120 mg/day oral prednisone or equivalent and, in the judgment of the investigator, expected to benefit from the addition of immunosuppressive therapy
* For women who are not postmenopausal (>/=12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two effective methods of contraception, including at least one method with a failure rate of less than (<) 1 percent (%) per year, during the treatment period and for at least 12 months after the last dose of study treatment

Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Barrier methods must always be supplemented with the use of a spermicide

Examples of contraceptive methods with a failure rate of < 1% per year (highly effective contraceptive methods) include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices

* For men (including those who have undergone a vasectomy): agreement to remain abstinent or use a condom during the treatment period and for at least 12 months after the last dose of study treatment and agreement to refrain from donating sperm during this same period

Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the participant

Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. In addition to male contraception, agreement to advise female partners of childbearing potential to use highly effective contraception during the study and for at least 12 months after the last dose of study treatment

* Agreement to avoid excessive exposure to sunlight during study participation
* Able to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

* Diagnosis of pemphigus foliaceus or evidence of paraneoplastic pemphigus or other non-PV autoimmune blistering disease
* History of a severe allergic or anaphylactic reaction to humanized or murine monoclonal antibodies, or known hypersensitivity to any component of rituximab
* Known hypersensitivity or contraindication to MMF, mycophenolic acid, polysorbate, or oral corticosteroids
* Lack of peripheral venous access
* Pregnant or lactating, or intending to become pregnant during the study

Women who are not postmenopausal (>/=12 months of non-therapy-induced amenorrhea) or surgically sterile must have two negative results with a sensitivity of >/=25 milli-international units per milliliter (mIU/mL): one from a serum pregnancy test at Day -8 to Day -10 of screening and another from a urine pregnancy test at Day 1 prior to randomization

* Participated in another interventional clinical trial within 28 days prior to randomization
* Use of any investigational agent within 28 days or 5 elimination half-lives prior to randomization (whichever is the longer)
* Significant cardiovascular or pulmonary disease (including obstructive pulmonary disease)
* Evidence of any new or uncontrolled concomitant disease that, in the investigator's judgment, would preclude participant participation, including but not limited to nervous system, renal, hepatic, endocrine, malignant, or gastrointestinal disorders
* Any concomitant condition that required treatment with oral or systemic corticosteroids within 12 weeks prior to randomization
* Treatment with intravenous (IV) immunoglobulin (Ig), plasmapheresis, or other similar procedure within 8 weeks prior to randomization
* Treatment with immunosuppressive medications (e.g., azathioprine, MMF) within 1 week prior to randomization
* Treatment with cyclophosphamide within 12 weeks prior to randomization
* History of or currently active primary or secondary immunodeficiency, including known history of HIV infection and other severe immunodeficiency blood disorders
* Known active infection of any kind (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV anti-infectives within 4 weeks prior to screening, or completion of oral anti-infectives within 2 weeks prior to randomization; entry into this study may be reconsidered once the infection has fully resolved
* History of or current cancer, including solid tumors, hematologic malignancies, and carcinoma in situ (except complete excision of basal cell of the skin and squamous cell carcinoma of the skin that have been treated or excised and cured)
* Currently active alcohol or drug abuse, or history of alcohol or drug abuse within 24 weeks prior to screening
* Major surgery within 4 weeks prior to randomization, excluding diagnostic surgery
* Treatment with rituximab or a B cell-targeted therapy (e.g., anti-cluster of differentiation [CD] 20 [CD20], anti CD22, or anti-B-lymphocyte stimulator [BLyS]) within 12 months prior to randomization
* Treatment with a live or attenuated vaccine within 28 days prior to randomization; it is recommended that a participant's vaccination record and the need for immunization prior to study entry be carefully investigated
* Evidence of abnormal liver enzymes or hematology laboratory values
* Positive test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) serology at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (68):
- United States (15):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona Medical Research Office, Tucson, Arizona
  - UC Davis Department of Dermatology, Sacramento, California
  - Univ of Calif-San Francisco, San Francisco, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital Dermatology, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - St Louis University Hospital, St Louis, Missouri
  - Uni of NY and Roswell Cancer, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest Baptist Hospital Center for Dermatology Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences Uni, Portland, Oregon
  - Penn University, Philadelphia, Pennsylvania
- Argentina (4):
  - Hospital Italiano, Buenos Aires
  - Hospital Luis Lagomaggiore, Mendoza
  - Hospital Austral, Pilar, Pcia de Buenos Aires
  - Centro de Investigaciones Médicas - CIM, San Juan Bautista
- Australia (2):
  - St George Hospital, Kogarah, New South Wales, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
- Brazil (3):
  - Faculdade de Medicina de Botucatu - Hospital das Clínicas, Botucatu, São Paulo
  - Santa Casa de São Paulo Hospital Central X, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Guildford Dermatology, Surrey, British Columbia
  - Lynde Institute for Dermatology, Markham, Ontario
- France (8):
  - Department of Dermatology Avicenne Hospital & University, Bobigny
  - CHU Hopitaux de Bordeaux, CHU Hopitaux de Bordeaux
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - Les Hospices Civils de Lyon Dermatologie inflammatoire et médecine interne, Lyon / Pierre Bénite
  - CHU de Reims, Reims
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
- Germany (7):
  - Klinik und Poliklinik für Dermatologie und Venerologie Universitätsklinikum Köln, Cologne
  - University Hospital for Dermatology, Dresden
  - Kompetenzzentrum Fragile Haut Klinik fur Dermatologie und Venerologie, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - University Hospital Schleswig-Holstein, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Hautklinik und Poliklinik, Mainz
  - University of Munster, Münster
- Israel (5):
  - HaEmek MC, Afula
  - Rambam Medical Centre; Dept. of Dermatology, Haifa
  - Rabin Medical Centre; Dept. of Dermatology, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Centre, Tel Aviv
- Italy (6):
  - Ambulatorio di Malattie Rare e Immunopatologia Cutanea, Florence, Lazio
  - Università di Parma Clinica Dermatologica, Parma, Lazio
  - U.O. Dermatologia Dipartimento Malattie Infettive Fondazione IRCCS Policlinico San Matteo, Pavia, Lazio
  - Centro Clinico per le genodermatosi Dipartimento di Dermatologia dell'Immacolata - IRCCS, Rome, Lazio
  - S.C. Dermatologia 2 - Ambulatorio Malattie Rare, Turin, Lazio
  - ASST DEGLI SPEDALI CIVILI DI BRESCIA; Clinica Dermatologica, Brescia, Lombardy
- Spain (4):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clínic. Barcelona, Barcelona
  - Hosp. G. U Gregorio Marañón, Madrid
  - Hospital de la Victoria, Málaga
- Turkey (Türkiye) (9):
  - Gülhane Military Medical Academy in Ankara, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Gaziantep University Medical Faculty Sahinbey Hospital, Gaziantep
  - Bezm-i Alem University Medical Faculty, Istanbul
  - Istanbul Uni Istanbul Medical Faculty, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Marmara Uni, Istanbul
  - Celal Bayar University Medical Faculty Hafsa Sultan Hospital, Manisa
  - Karadeniz Teknik Üniversitesi Tıp Fakültesi Farabi Hastanesi, Trabzon
- Ukraine (2):
  - Dnipropetrovsk State Medical Academy, Dnipropterovsk
  - Territorial Medical Association "Dermatovenerologia", Kyiv

REFERENCES:
- [Derived] Werth VP, Joly P, Mimouni D, Maverakis E, Caux F, Lehane P, Gearhart L, Kapre A, Pordeli P, Chen DM; PEMPHIX Study Group. Rituximab versus Mycophenolate Mofetil in Patients with Pemphigus Vulgaris. N Engl J Med. 2021 Jun 17;384(24):2295-2305. doi: 10.1056/NEJMoa2028564. Epub 2021 May 19. PMID 34097368

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab (RTX): Participants received rituximab by IV infusion on Days 1 and 15 with repeat administration on Days 168 and 182 provided specific safety criteria had been met. Participants also received MMF matching placebo orally twice daily (every 12 hours, Q12H) from Day 1 to Week 52. Participants who withdrew from the treatment period or who completed the total 52-week treatment period entered the safety follow up (SFU) period, and they were observed for 1 year and did not receive any further study treatment.
- Mycophenolate Mofetil (MMF): Participants received Mycophenolate Mofetil (MMF) orally twice daily (every 12 hours, Q12H) from Day 1 to Week 52. Participants also received rituximab matching placebo by intravenous (IV) infusion on Days 1 and 15 with repeat administration on Days 168 and 182 provided specific safety criteria had been met. Participants who withdrew from the treatment period or who completed the total 52-week treatment period entered the safety follow up (SFU) period, and they were observed for 1 year and did not receive any further study treatment.
Period: Treatment Period
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Started | 67 | 68
Completed (Completed the 52-week treatment period and entered safety follow up (SFU)) | 66 | 58
Not Completed | 1 | 10
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Non-compliance with study drug | 0 | 1
Period: Safety Follow-up (SFU)
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Started | 66 | 58
Completed | 59 | 53
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Treated by not accepted treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF) | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.66 (12.98) | 46.34 (13.08) | 48.48 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 32 | 30 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 21 | 34
  Not Hispanic or Latino | 45 | 41 | 86
  Not Stated | 8 | 5 | 13
  Unknown | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Black or African American | 1 | 2 | 3
  White | 49 | 51 | 100
  Unknown | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (Excluding Telemedicine [TM] Participants) Who Achieved Sustained Complete Remission, Evaluated by the Pemphigus Disease Area Index (PDAI) Activity Score
Time Frame: From Baseline up to 52 Weeks (up to clinical cut-off date (CCOD) of 28 November 2018)
Population: The modified intent-to-treat (mITT) population included participants in the ITT population (all randomized participants who received any part of an infusion of study drug or oral administration of study drug), excluding the 10 telemedicine (TM) participants. This population was used in the analyses of efficacy outcomes.
Measure: Number; unit: Percentage of Participants
Groups:
- Rituximab (RTX): Participants received rituximab by IV infusion on Days 1 and 15 with repeat administration on Days 168 and 182 provided specific safety criteria had been met. Participants also received MMF matching placebo orally twice daily (every 12 hours, Q12H) from Day 1 to Week 52.
- Mycophenolate Mofetil (MMF): Participants received Mycophenolate Mofetil (MMF) orally twice daily (every 12 hours, Q12H) from Day 1 to Week 52. Participants also received rituximab matching placebo by intravenous (IV) infusion on Days 1 and 15 with repeat administration on Days 168 and 182 provided specific safety criteria had been met.
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 62 | 63
Percentage of Participants | 40.3 | 9.5
Statistical Analysis 1: Comparison: Rituximab (RTX) vs Mycophenolate Mofetil (MMF); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The analysis was stratified by the stratification factors applied at randomization; Difference in proportion = 30.80, 95% CI 2-sided [14.70 to 45.15]

2. Secondary Outcome: Cumulative Oral Corticosteroid Dose
Time Frame: From Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: The mITT population included participants in the ITT population (all randomized participants who received any part of an infusion of study drug or oral administration of study drug), excluding the 10 TM participants. This population was used in the analyses of efficacy outcomes.
Measure: Median (Inter-Quartile Range); unit: milligram (mg)
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 62 | 63
milligram (mg) | 2775.00 [2146.88 to 3610.00] | 4005.00 [2662.50 to 5815.00]
Statistical Analysis 1: Comparison: Rituximab (RTX) vs Mycophenolate Mofetil (MMF); Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Number of Protocol Defined Disease Flares
Description: Disease flare is defined as appearance of three or more new lesions a month that do not heal spontaneously within 1 week, or by the extension of established lesions, in a participant who has achieved disease control.
Time Frame: From Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: as for outcome 2
Measure: Number; unit: Number of Flares
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 62 | 63
Number of Flares | 6 | 44
Statistical Analysis 1: Comparison: Rituximab (RTX) vs Mycophenolate Mofetil (MMF); Test type: Superiority; p < 0.0001, Negative Binominal Regression — The model was adjusted for the following covariates in addition to log (each participant's duration in study) as an offset: treatment, region, duration of illness, baseline PDAI activity score, and baseline prednisone dose; Adjusted Rate Ratio = 0.12, 95% CI 2-sided [0.05 to 0.29]

4. Secondary Outcome: Time to Initial Sustained Complete Remission
Time Frame: From Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 62 | 63
Weeks | NA [32.1 to NA] — The median is not estimable due to limited number of events | NA [NA to NA] — The median is not estimable due to limited number of events
Statistical Analysis 1: Comparison: Rituximab (RTX) vs Mycophenolate Mofetil (MMF); Test type: Superiority; p = 0.0003, Log Rank — P-value is from a stratified log-rank test used to test the time to first disease flare between the RTX and MMF treatment arms over the 52-week treatment period, adjusting for the stratification factors applied at randomization; Hazard Ratio (HR) = 4.83, 95% CI 2-sided [1.97 to 11.81]

5. Secondary Outcome: Time to Protocol Defined Disease Flare
Description: Disease flare is defined as the appearance of three or more new lesions a month that do not heal spontaneously within 1 week or by the extension of established lesions in a participant who has achieved disease control.
Time Frame: From Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 62 | 63
Weeks | NA [NA to NA] — The median is not estimable due to limited number of events | NA [36.9 to NA] — The median is not estimable due to limited number of events
Statistical Analysis 1: Comparison: Rituximab (RTX) vs Mycophenolate Mofetil (MMF); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.15, 95% CI 2-sided [0.06 to 0.39]

6. Secondary Outcome: Change in Health-Related Quality of Life (HRQoL), as Measured by the Dermatology Life Quality Index (DLQI) Score
Description: Total DLQI scores range from 0 to 30 with higher DLQI scores reflecting greater impairment in a participant's health-related quality of life. The DLQI score is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The measure type mean is the estimated mean from adjusted MMRM.
Time Frame: From Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: The mITT population included participants in the ITT population (all randomized participants who received any part of an infusion of study drug or oral administration of study drug), excluding the 10 TM participants. This population was used in the analyses of efficacy outcomes. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 62 | 63
Scores on a Scale
  Baseline: number analyzed (Participants) | 57 | 58
  Baseline | 10.14 (7.89) | 11.09 (8.52)
  Week 52: number analyzed (Participants) | 45 | 27
  Week 52 | -8.874 (0.532) | -6.002 (0.662)
Statistical Analysis 1: Comparison: Rituximab (RTX) vs Mycophenolate Mofetil (MMF); Test type: Superiority; p = 0.0012, Mixed Model Repeated Measures — P-value is from Mixed Model Repeated Measures (MMRM) with unstructured covariance matrix, adjusting for treatment, region, duration of illness, baseline DLQI score, visit, and an interaction terms for visit × baseline DLQI score and visit × treatment; Difference in Estimated Means = -2.872, 95% CI 2-sided [-4.577 to -1.167]

7. Secondary Outcome: Percentage of Participants With Adverse Events, Serious Adverse Events, and Corticosteroid-Related Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant to whom a medicinal product is administered and which does not necessarily have a causal relationship with this treatment. A serious adverse event is an adverse event that results in death or is life-threatening or requires/prolongs hospitalization or results in persistent/significant disability/incapacity or congenital abnormality/birth defect. Adverse events of Grade 3 of higher are severe and life-threatening adverse events CS-related adverse events - causality as determined by the investigator.
Time Frame: Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: The safety population included all participants who were randomized and received any part of an infusion of study drug or oral administration of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 67 | 68
Percentage of Participants
  Participants with AE | 85.1 | 88.2
  Participants with SAE | 22.4 | 14.7
  Participants with Corticosteroid (CS)-Related AE | 34.3 | 38.2
  Participants with CS-Related AE Grade 3 or higher | 1.5 | 7.4

8. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA)
Description: Participants with treatment-induced and treatment-enhanced anti-drug antibodies. The clinical relevance of anti-rituximab antibody formation in RITUXAN treated pemphigus vulgaris (PV) participants is unclear.
Time Frame: Baseline up to 52 Weeks (up to CCOD of 28 November 2018)
Population: The safety population (all participants who were randomized and received any part of an infusion of study drug), only participants for whom data were collected are included in the analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab (RTX)
Number analyzed (Participants) | 67
Percentage of Participants | 31.7

9. Secondary Outcome: Percentage of Participants With Immunoglobulin (Ig) Levels Below Lower Limit of Normal (LLN)
Time Frame: Baseline; Weeks 16, 24, 40 and 52; (end of treatment: up to Week 52) (up to CCOD of 28 November 2018)
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 67 | 68
Percentage of Participants
  Baseline (IgA) | 0 | 0
  Week 16 (IgA) | 0 | 1.8
  Week 24 (IgA) | 1.7 | 2.2
  Week 40 (IgA) | 0 | 2.7
  Week 52 (IgA) | 0 | 3.6
  Baseline (IgG) | 6.1 | 6.0
  Week 16 (IgG) | 9.8 | 1.8
  Week 24 (IgG) | 3.4 | 2.2
  Week 40 (IgG) | 3.5 | 0
  Week 52 (IgG) | 4.3 | 0
  Baseline (IgM) | 7.6 | 11.9
  Week 16 (IgM) | 24.6 | 23.2
  Week 24 (IgM) | 27.1 | 28.3
  Week 40 (IgM) | 29.8 | 24.3
  Week 52 (IgM) | 29.8 | 28.6

ADVERSE EVENTS:
Time Frame: Treatment Period: From Baseline up to Week 52 (up to CCOD of 28 November 2018) Safety Follow-up Period: Approximately 1 year (up to CCOD of 29 October 2019)
Description: The safety population included all participants who were randomized and received any part of an infusion of study drug or oral administration of study drug. Participants who received the incorrect therapy from that assigned were summarized according to the therapy actually received. This population was used for the analyses of safety outcomes. Only serious adverse events and all infectious adverse events, irrespective of causality, were reported in the SFU period.
Groups:
- RTX Safety Follow-up: Participants, who received RTX in the treatment period, and either withdrew from the treatment period or completed the total 52-week treatment period, entered the SFU period. Participants were observed for 1 year and did not receive any further study treatment.
- MMF Safety Follow-up: Participants, who received MMF in the treatment period, and either withdrew from the treatment period or completed the total 52-week treatment period, entered the SFU period. Participants were observed for 1 year and did not receive any further study treatment.
Arm/Group | Rituximab (RTX) | Mycophenolate Mofetil (MMF) | RTX Safety Follow-up | MMF Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 0/67 | 1/68 | 0/66 | 0/58
Serious Adverse Events (participants affected / at risk) | 15/67 | 10/68 | 4/66 | 1/58
Other Adverse Events (participants affected / at risk) | 42/67 | 41/68 | 2/66 | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (RTX) (N=67) | Mycophenolate Mofetil (MMF) (N=68) | RTX Safety Follow-up (N=66) | MMF Safety Follow-up (N=58)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (RTX) (N=67) | Mycophenolate Mofetil (MMF) (N=68) | RTX Safety Follow-up (N=66) | MMF Safety Follow-up (N=58)
LYMPHOPENIA (Blood and lymphatic system disorders) | 8 (14) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (5) | 10 (11) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (4) | 4 (4) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 4 (5) | 4 (4) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 5 (8) | 3 (3) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 6 (8) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 6 (8) | 8 (12) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 6 (8) | 6 (6) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (9) | 5 (6) | 2 (2) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 12 (19) | 5 (6) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 10 (17) | 6 (7) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02383589/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT02383589/SAP_003.pdf